CLINICAL TRIAL: NCT02895477
Title: Quest Sound Recover (SR2) vs. Venture SR2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Sonova2016_10
Record Dates: First submitted 2016-08-29; First posted 2016-09-09 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss | interventions — Hearing Aids

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Intervention group (Experimental): Hearing aid
  Interventions: Device: hearing aid
- Test group (Experimental): Hearing aid
  Interventions: Device: hearing aid

INTERVENTIONS:
Device: hearing aid

SUMMARY:
Goal of this study is to determine the benefit of an improved feature on a new hearing aid platform.

To investigate the improvements of this feature is compared on a new and older hearing aid platform. The obtained results will be used for future improvement for this feature. This feature should improve the speech understanding and speech recognition of the hearing aid user.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature (Appendix Informed Consent Form)
* Ability to fill in a question conscientious
* Healthy outer ear (w/o previous surgical procedures)
* Sensorineural symmetric hearing loss (HL)
* N4 to N7 (degree of HL)

Exclusion Criteria:

* Contraindications to the MD in this study, e.g. known hypersensitivity or allergy to the investigational product,
* Limited mobility and not in the position to attend weekly appointments
* Limited ability to describe listening impressions/experiences and the use of the hearing aid
* Inability to produce a reliable hearing test result when pure tone audiometry is attempted by the audiologist
* Massively limited dexterity
* Known Psychological problems
* Central hearing problems

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-07; Primary Completion 2016-12 (Actual); Study Completion 2017-01-20 (Actual)

PRIMARY OUTCOMES:
Functional gain | after 2 weeks
  Functional gain is to measure the aided threshold (in dB hearing level [HL]) in free field via loudspeaker.
Phoneme Perception Test | after 2
  Change of Detection thresholds after 4 weeks hearing instrument wearing time
Functional gain | after 8 weeks
  Functional gain is to measure the aided threshold (in dB hearing level [HL]) in free field via loudspeaker.
Phoneme Perception Test | after 8 weeks
  Change of detection thresholds after 4 weeks hearing instrument wearing time

SECONDARY OUTCOMES:
sound quality ratings | after 6 and 12 weeks
questionnaires | after 2, 6, 8 and 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Sonova AG, Stäfa, Canton of Zurich, Switzerland